CLINICAL TRIAL: NCT06191510
Title: Effect of Healing Xenogenic Biomaterial Exposed to the Oral Environment in Humans
Brief Title: Xenogenic Bone Intentionally Left Exposed
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: São Paulo State University (Other); Universidade Federal de Sergipe (Other)
Responsible Party: Principal Investigator, Arthur Belem Novaes Jr, Phd, Ms, DDs. Chairman of Periodontolgy, University of Sao Paulo
Other Study IDs: CAAE: 21305419.1.0000.5419
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Soft Tissue; Dental Implants; Healing Wound
Keywords: Molar site; Alveolar Bone Loss; Tissue Conditioning, Dental; Biomaterials
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Biocompatible Materials

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental Group: The aim of this study is to assess the effectiveness of usage of xenogeneic bone intentionally left exposed to the oral environment after immediate implant placement in preserving keratinized mucosa and the alveolar ridge height and width preservation, without compromising the healing process.
  Interventions: Procedure: Bio-Oss Exposed
- Control group: The aim of this study is to evaluate whether the use of collagen matrix has benefits when compared to xenogeneic bone intentionally left exposed to the oral environment after immediate implant placement.
  Interventions: Procedure: Mucograft Exposed

INTERVENTIONS:
Procedure: Bio-Oss Exposed — Molar extraction with a flapless approach and immediate implant installation, filling the gap with deproteinized bovine bone mineral (Geistlich Bio-Oss) and left exposed to the oral environment.
  Other Names: Immediate Implant Placement Associated with biomaterials
  Groups: Experimental Group
Procedure: Mucograft Exposed — Molar extraction with a flapless approach and immediate implant installation, filling the gap with deproteinized bovine bone mineral (Bio-Oss; Geistlich) and covered by a collagen matrix (Mucograft; Geistlich).
  Other Names: Immediate Implant Placement Associated with biomaterials
  Groups: Control group

SUMMARY:
The goal of this clinical trial is to compare, the effect of letting the xenogeneic bone graft exposed to the oral environment or seal off the graft with a collagen matrix. Them main questions it aims to answer are:

* The enhancement of soft tissue healing during the initial phases following immediate implant placement.
* The secondary aim is to evaluate the dimensional alterations in hard tissues at immediately placed implants and different biomaterial protocol.

It were selected patients with indication of flapless extraction in posterior teeth, which was placed immediate implant (n=28) and gap filling with deproteinized bovine bone mineral (Geistlich Bio-Oss®). In this study, participants were stratified into two randomized blocks, each corresponding to a distinct surgical technique: left exposed the graft to the oral environment or coverage with a collagen matrix (Geistlich Mucograft®).

* Previously the extraction was performed the measurement of the keratinized gingiva, and after 04 months of implant placement.
* The soft tissue healing was evaluated on days 02, 07, 30 days; by means of a blue-stained solution (methylene blue 0.05%) and standardized photograph.
* In the same date from different healing times it was performed immunoenzymatic analysis of the levels of VEGF (vascular endothelial growth factor), IL-1β (interleukin-1β) and FGF2 (fibroblast growth factor 2).
* It was also be performed cone beam computed tomography images quantifying the soft and hard tissues thickness of the facial and lingual bone wall. The clinical trial examiner was blinded during the study period.

DETAILED DESCRIPTION:
The present study aimed to evaluate molecular, histologically and tomographic soft and hard tissue parameters of tissue healing in immediate placement of dental implant and gap filling with Bio-Oss covered (control group), or not (test group) with Mucograft. he hypothesis was that both the test group and the control group would have great results in alveolar preservation.

The implant function successful does not reach the patients and clinicians aesthetic demands, as well the approach and integrity of hard and soft tissue structures, which are compromised by physiological and structural changes after the dental extraction, are challenge in the implant treatment (Chappuis et al., 2017). The alveolar process is tooth dependent, and the dimensional alterations of the alveolar ridge that occurred following tooth extraction in a thin bone phenotype (< 1 mm) is inherent in the healing process, but can be minimized by alveolar preservation (Ten Heggeler et al., 2011; Jung et al., 2013; Sculean et al., 2014; Chappuis et al., 2017; Jung et al., 2018). A systematic review revealed 2.6 to 4.5 mm in width bone loss and 0.4 to 3.9 mm vertically in non-molar regions following tooth extraction (Ten Heggeler et al., 2011). This loss could be reduced from 43.3% to 18.1% by using bone grafts and covering the alveolus with free gingival grafts in a 6-month follow-up (Jung et al., 2018). Several studies focused on bone healing parameters, placing bone substitute materials in alveolar sockets to reduce resorption after tooth extractions. However, soft tissue healing after extraction received little attention in clinical research.

The average and standard deviation of group 1 were 4 and 0.8, respectively, and for group 2, they were 5 and 1. To verify the variation in amount of keratinized tissue considered clinically relevant and different between groups was calculated (GPower 3.1). A sample for a total of 28 immediate implant placement, being equivalent to each group (14 for group 1 and 14 for group 2), taking into account a significance level of 5%, 80% test power and average difference of 1.0 mm between the groups and standard deviation of 20%. The study was a Randomized Controlled Clinical Trial, with clinical procedures conducted by an experienced dentist, and the examiner analyzing the entire trial blinded during the study period.

The selection included patients requiring extraction of at least one posterior tooth due to caries, endodontic complications, periodontitis, orthodontic and prosthetic reasons. Only healthy patients with adequate oral hygiene (bleeding on probing ≤ 10% and plaque), primary stability of at least 35N after implant placement. The exclusion criteria were: age < 18 years, smoking; smoking more than 10 cigarettes per day; presence of relevant medical conditions: diabetes mellitus, unstable or potentially fatal conditions or requiring antibiotic prophylaxis and drug medication that influence bone metabolism; pregnant or lactating women; radiotherapy or chemotherapy for malignancy in the last 5 years; history of autoimmune disease; presence of acute periodontal or periapical pathology; and history of drugs or elitist. . Patients were invited to participate after ethical committee approval, and randomization into blocks was done through an online application.

A comprehensive periodontal examination was conducted before any surgical procedure. Keratinized gingiva width was evaluated using a periodontal probe at the facial level, measuring the distance from the muco-gingival junction and gingival margin before extraction and after 4 months at implant placement. Flapless tooth extraction was performed in the least traumatic way, and dental implants (Straumann SLActive) were immediately placed. The buccal gap was filled with xenogeneic deproteinized bovine bone (Geistlich Bio-Oss®). In the study group, bone grafting was exposed with flap healing by second intention, while in the control group the collagen matrix (Geistlich Mucograft®) was pulled over the healing cap. Standard postoperative instructions were given, and Amoxicillin 875 mg (every 12 hours for 11 days) was prescribed 24 hours before the surgical intervention, along with analgesics every 6 hours for 3 days.

At each follow-up visit (02, 07, 30 days) the surgical area was stained with methylene blue (0,05%) to check for surface epithelialization. The lesions are stained so that they are easily distinguishable. This solution has been suggested to identification of minor areas lacking epithelium (Kohale et al., 2018). Tthe chosen dates corresponded to the stages of tissue healing: initial (0 - 3 days), revascularization (4-11 days), and maturation of tissue (11-42 days). Clinical measurements recorded on days 2, 7, and 30 postoperatively were photographed by occlusal view, and epithelium scores were evaluated, classified as follows (Jung et al., 2018): Grade 1: non-existent; Grade 2: covering less than one-quarter of the wound surface; Grade 3: covering less than half the wound surface; Grade 4: covering more than three-quarters of the wound surface; and Grade 5: normal or complete covering of the wound.

The regulation of anti-inflammatory cytokines VEGF and IL-10, and pro-inflammatory IL-1β and TNF-α (tumor necrosis factor-α) are key factors in wound healing, in which the increase of these latter cytokines are indicative of delayed healing. VEGF is a vascular endothelial growth factor, being one of the main stimulators of the formation of new blood vessels (Sculean et al., 2014). Thus, in the immunoenzymatic analysis, the levels of VEGF, IL-1β and FGF2 were evaluated. Fluid samples from the wound were obtained by means of a stick with sterile swab, slow rolling movements, edge-to-edge, after little irrigation with sterile saline solution. Then the the swabs were placed in 2 mL microtubes and samples were frozen at -80° C until analyzed. Immunoenzymatic analysis was conducted to evaluate the levels of VEGF, IL-1β, and FGF2 in fluid samples obtained from the wound. Commercial kits and Luminex/MAGpix technique were used for quantitative cytokine levels determination from a fifth-degree polynomial curve using the xPONENT Software® (Luminex Corporation, Austin, TX, EUA).

For the evaluation of bone thickness and soft tissues, cone beam computed tomography (CBCT) imaging was used. Patients used mouth retractors and were instructed to stay with the tongue retracted, directed to the palate, and it was possible to distinguish the soft tissues of the lips, cheeks and gums. The CBCT were acquired with the iCAT software on a computer. A scan was taken of the maxilla (scan dimensions of 6x17 cm) for 40 seconds with the following setting of the iCAT-voxel size: 0.2 mm; gray scale: 14 bits; focal spot: 0.5 mm; image detector: amorphous silicone flat panel; image acquisition: single 360° rotation. The scan was performed after surgery and in the fourth following month, evaluating bone thickness and gingival tissue. An open software package (Slicer 3.6. www.slicer.org) was used for the overlap of the original DICOM data of the two tomographies, evaluating bone thickness and gingival tissue. Thus, the two image sets were aligned and checked manually for perfect match (Jung et al., 2013). Reference lines were drawn based on the most apical point of the extraction outlet and the apex of the implant. The vertical reference line was drawn at the center of the extraction outlet crossing the apical reference point. The horizontal reference line was drawn perpendicularly to the vertical line crossing the apical reference point. Standardized measurements evaluated horizontal bone thickness, both vestibular and lingual, from traces delimited 2 mm below the implant machined collar (reference line - RL), RL, -2, -1 and 0 mm above this line. Soft tissue thickness was evaluated at baseline and alterations after 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (≥18 years-old) exhibiting good oral hygiene,
* Hopeless molar teeth with an intact buccal socket wall,
* Sufficient apical bone allowing for immediate implant placement.

Exclusion Criteria:

* Individuals with systemic diseases that are unstable,
* Uncontrolled metabolic conditions,
* Daily smoking habit of ≥10 cigarettes,
* Those who have received antibiotic drugs or corticosteroids within the past 3 months, or are currently on medications that impact bone healing, such as bisphosphonates,
* Patients with a past history of chemotherapy or radiation therapy in the oral and maxillofacial region.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hopeless molar teeth who are scheduled for immediate implant placement in this area, in the researcher's town.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Keratinized Mucosa Width | before extraction, after 1-2 months post implant placement, and after the emergence contour of a prosthesis (up to 4 months).
  The keratinized mucosa width was evaluated using a periodontal probe at the facial level before extraction and after 4 months at the implant placement.

SECONDARY OUTCOMES:
Cone Beam Computed Tomographs Measurements | Baseline; after 4 months
  To assess in tooth, prior to extraction, mucosal thickness and changes in alveolar ridge height and width, a cone beam computed tomographs (CBCT) images were obtained under consistent conditions. All radiographic measurements and analyses were conducted both at baseline (after the implant placement) and after 4 months.

OTHER OUTCOMES:
Clinical Assessment of Epithelialization | 2 day, 1 week, and 1 month after the implant placement
  Clinical measurements were recorded at 2 day, 1 week, and 1 month postoperatively and assessed as scores of epithelialization, graded as follows:
  * Grade 1: non-existent
  * Grade 2: covering less than one-quarter of the wound surface
  * Grade 3: covering less than half the wound surface
  * Grade 4: covering more than three-quarters of the wound surface
  * Grade 5: normal or complete covering of the wound.
Serum levels of cytokines | 2 day, 1 week, and 1 month after the implant placement
  The cytokine content of each sample (evaluated on days 02, 07, 30 days of healing) was measured by multiplex assay. The cytokines analyzed were VEGF, IL-1β and FGF2.

CONTACTS AND LOCATIONS:
Overall Officials: Valessa F Carvalho, PhD student, Principal Investigator — School of Dentistry of Ribeirão Preto
Locations (1):
- School of Dentistry of Ribeirão Preto - University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No